CLINICAL TRIAL: NCT06947005
Title: The Effect of Serious Game and Video-Assisted Education on Nursing Students' Psychomotor Skill Development, Perception of Clinical Stress, Satisfaction and Self-Confidence in Learning
Brief Title: The Effect of Serious Game and Video-Assisted Education on Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Hakime Aslan, Principal Investigator, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Tülay Çetkin
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Nursing Students
Keywords: Nursing students; Serious Game; Psychomotor Skills; Stress; Video-Assisted Learning

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): Serious game group
  Interventions: Behavioral: Intervention 1
- Intervention 2 (Experimental): Video asisted learning group
  Interventions: Behavioral: Intervention 2
- Control group (No Intervention): Control

INTERVENTIONS:
Behavioral: Intervention 1 — The students in the serious game group were asked to download the drug applications serious game to their phones. They were asked to play the game for two weeks. The students continued to play the game at any time and as often as they wanted until they won at least one gold medal for each application. At the end of the 2nd week, a questionnaire form and VAS scale were applied to the students to evaluate the post-test data and their satisfaction levels with the game. The collected data were analysed to understand the different dimensions of game satisfaction and to assess overall satisfaction levels.
  Other Names: Serious game
  Arms: Intervention
Behavioral: Intervention 2 — A WhatsApp group was established to maintain communication with the students in the video-supported education group. After the pre-test data were collected, the students were introduced to the ed-puzzle web page where they could watch the application videos and were asked to register to the system. No fee was paid to register to the ed-puzzle web page. Students were given the opportunity to watch the videos on the ed-puzzle web page for 2 weeks and answer the questions. Each student was allowed to watch the videos at least once until they answered all the questions correctly. The number of videos watched was monitored by the researcher. At the end of the 2nd week, post-test data were collected from the students.
  Other Names: Video assited learning
  Arms: Intervention 2

SUMMARY:
Aim: This study was conducted to evaluate the effect of a serious game and video-assisted training program developed for parenteral drug administration education on nursing students' psychomotor skill development, perception of clinical stress, satisfaction, and self-confidence in learning.

Material and Method: The study was carried out as a randomized controlled experimental research design between June 2023 and April 2025 at the Faculty of Nursing, İnönü University. All students enrolled in the Nursing Department during the Spring Semester of the 2023-2024 academic year constituted the study population. The sample consisted of 99 students (33 in the serious game group, 33 in the video group, and 33 in the control group), determined by power analysis. Data were collected using the "Psychomotor Skills Evaluation Checklists," the "Perceived Stress Scale for Nursing Students," and the "Student Satisfaction and Self-Confidence in Learning Scale."

DETAILED DESCRIPTION:
Serious games help to develop participants' problem solving, critical thinking and communication skills, while enriching the learning experience. Serious gaming is a learning-first approach that mimics reality using virtual simulation. These games can be used to optimise the acquisition of clinical skills, stimulate student motivation by completing the simulation and allow teachers to assess students' progress.Video-assisted learning provides learners with a visual tool that facilitates the understanding of abilities and skills. It is often used to illustrate how a teacher or expert addresses a topic, process or skill. The content can then be followed, learnt and applied by learners. In this study, both methods were evaluated together and their effects on the development of nursing students' competencies for parenteral drug adminstrantion practices were evaluated

ELIGIBILITY:
Inclusion Criteria:

* Being a 1st year nursing student,
* Receiving training on parenteral drug applications for the first time,
* Not having any physical disabilities related to vision, hearing and motor skills,
* Having a smart mobile phone with Android/IOS operating system, and
* Volunteering to participate in the study.

Exclusion Criteria:

* Students who made vertical transfer to the department with DGS because they may have taken the subject of parenteral drug applications in an associate degree programme before,
* Students who did not have a smart mobile phone with Android / IOS operating system and
* Students who did not volunteer to participate in the study were excluded from the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Effect of Student Satisfaction and Confidence in Learning | 2 weeks later
  For the pre-test data, the students were given the "Individual Introduction Form" and the "Student Satisfaction and Confidence in Learning Scale" and asked to fill them in.
  At the end of the 2nd week, the "Student Satisfaction and Confidence in Learning Scale" was applied again to evaluate the satisfaction and self-confidence of the students who received training with different teaching methods for 2 weeks.
  The Student Satisfaction and Confidence in Learning Scale was developed to measure the satisfaction and self-confidence of nursing students who experience learning with simulation method. The Turkish validity and reliability study of the scale was conducted by Karaçay and Kaya in 2015. The scale consists of a total of 13 items and 2 sub-dimensions (satisfaction with learning and self-confidence). A score between 13-65 can be obtained from the scale developed in 5-point Likert type. A high score on the scale indicates high 'student satisfaction and self-confidence'.
Effect of Perceived Stress | 2 weeks later
  For the pre-test data, the students were given the "Perceived Stress Scale for Nursing Students" and asked to fill them in.
  At the end of the 2nd week, the "Perceived Stress Scale for Nursing Students" was applied again to evaluate the stress of the students who received training with different teaching methods for 2 weeks. The Perceived Stress Scale for Nursing Students was developed to determine the level and type of stress perceived by nursing students in clinical practice. Turkish validity and reliability study was conducted in 2015. The scale consists of a total of 29 items and 6 sub-dimensions. A score between 0-116 can be obtained from the scale developed in 5-point Likert type. A high score on the scale indicates a high degree of stress.
Effect of psychomotor skills | 2 weeks later
  In order to evaluate the psychomotor skill level of the students in the groups, the researcher and the independent observer evaluated the drug administration skills of each student individually and filled out the 'Psychomotor Skill Assessment Checklists for Drug administration'. The skill evaluation process of each student lasted 10-15 minutes.
  Skill checklists were developed to evaluate the skill performance of students on urinary system applications. Skill checklists are step-by-step checklists showing the skills expected to be performed by students and were prepared by reviewing the relevant current literature.

CONTACTS AND LOCATIONS:
Overall Officials: Hakime Aslan, Study Director — Faculty of Nursing
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)